CLINICAL TRIAL: NCT02930343
Title: Comparison of Sulfasalazine Versus Leflunomide Based Combination Disease Modifying Anti-rheumatic Drug Therapy (DMARD) in Patients With Rheumatoid Arthritis Failing Methotrexate Monotherapy : A Randomized Control Trial
Brief Title: Comparison of Disease Modifying Antirheumatic Drugs Therapy in Patients With RA Failing Methotrexate Monotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to time constraints, the study was halted prematurely
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Dr. Vir Singh Negi, Professor and head of the department, Department of Clinical Immunology, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIP/IEC/2016/27/893
Record Dates: First submitted 2016-09-13; First posted 2016-10-12 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Leflunomide; Hydroxychloroquine; Prednisolone; Steroids; Glucocorticoids; Folic Acid; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1- MTX+LEF+HCQ (Active Comparator): Active Comparator: Combination of Methotrexate (up to 25 mg per week), Leflunomide (20 mg once a day) and Hydroxychloroquine (200-400 mg once at night). All drugs are to be taken orally. Duration of therapy is for 3 months. All patients will receive folic acid (5 mg twice a week) along with methotrexate. Low dose prednisolone (weeks 1-2: 7.5 mg/day, weeks 2-4: 5 mg/day, weeks 4-6: 5 mg on alternate day and then stop) will be given as bridging therapy.
  Interventions: Drug: Methotrexate; Drug: Leflunomide; Drug: Hydroxychloroquine; Drug: Prednisolone; Drug: Folic Acid
- group 2- MTX+SSZ+HCQ (Active Comparator): Combination of Methotrexate (up to 25 mg per week), Sulfasalazine (2g per day) and Hydroxychloroquine (200-400 mg once at night). All drugs are to be taken orally. Duration of therapy is for 3 months. All patients will receive folic acid (5 mg twice a week) along with methotrexate. Low dose prednisolone (weeks 1-2: 7.5 mg/day, weeks 2-4: 5 mg/day, weeks 4-6: 5 mg on alternate day and then stop) will be given as bridging therapy.
  Interventions: Drug: Methotrexate; Drug: Hydroxychloroquine; Drug: Prednisolone; Drug: Folic Acid; Drug: Sulfasalazine

INTERVENTIONS:
Drug: Methotrexate — Methotrexate, a structural analogue of folic acid, can be administered orally or parenterally to treat a variety of rheumatic diseases
  Other Names: folitrax, MTX
Drug: Leflunomide — Leflunomide inhibits pyrimidine synthesis, resulting in blockade of T-cell proliferation. Leflunomide is used in patients with moderate to severe active rheumatoid arthritis with early or late disease
  Other Names: Arava, Lefno, LEF
  Arms: group 1- MTX+LEF+HCQ
Drug: Hydroxychloroquine — Hydroxychloroquine (HCQ) is a well-tolerated DMARD that is commonly used in combination therapy regimens for RA. HCQ is more commonly used than chloroquine.
  Other Names: HCQ
Drug: Prednisolone — Low dose prednisolone (weeks 1-2: 7.5 mg/day, weeks 2-4: 5 mg/day, weeks 4-6: 5 mg on alternate day and then stop)
  Other Names: Steroids, Glucocorticoids
Drug: Folic Acid — Folic acid is to be given to all patients receiving methotrexate at a dose of 5 mg twice a week.
  Other Names: Folvite
Drug: Sulfasalazine — 5-aminosalicylic acid (5-ASA) is the active component of sulfasalazine; the specific mechanism of action of 5-ASA is unknown; however, it is thought that it modulates local chemical mediators of the inflammatory response, especially leukotrienes, and is also postulated to be a free radical scavenger or an inhibitor of tumor necrosis factor (TNF)
  Other Names: Saaz, SSZ
  Arms: group 2- MTX+SSZ+HCQ

SUMMARY:
RA (Rheuatoid arthritis) is a multisystem disease that mainly involves joints resulting in destructive arthritis if not treated rapidly. Inspite of various advances in field of early diagnosis and treatment of RA, there is still a need for better understanding of the efficacy and safety of various combinations of conventional DMARDS, and to rank them in order accordingly, so as to give a clearer vision for further management of RA once MTX monotherapy fails, so as to achieve remission as soon as possible. The study will be conducted at the Department of Clinical Immunology, JIPMER (Jawaharlal Institute of Postgraduate Medical Education & Research). patients who fail methotrexate monotherapy will be randomised to 2 treatment arms - either a combination of Sulfasalazine (SSZ), Hydroxychloroquine (HCQ) and Methotrexate (MTX) or Leflunomide (LEF), Hydroxychloroquine (HCQ) and Methotrexate (MTX)

DETAILED DESCRIPTION:
Patients aged ≥18 years, fulfilling the 2010 ACR EULAR criteria for RA (symptom duration less than two years) , having more than 4 joints involved & having moderate to severe disease activity (DAS28≥3.2) will be invited to participate. After providing written informed consent, eligible patients will be first started on MTX monotherapy & only patients who have persistant moderate disease activity (DAS28 ESR > 3.2) will be randomized into two groups. Block randomization will be done to generate random allocation sequence

Group 1 - will receive MTX+LEF+HCQ Group 2- will receive MTX+SSZ+HCQ

DMARD dosages used are: MTX 25 mg/week orally (dosage after 6 weeks),SSZ 2g/d (after 4 weeks) LEF 20 mg/day (dosage after 2 weeks) and HCQ 200 mg/day. Glucocorticoids will be given in an oral tapering scheme. All patients will be prescribed folic acid (10 mg/week) during MTX prescription.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years satisfying ACR-EULAR criteria for RA

1. Polyarthritis (>4 joints)
2. Disease duration of less than 2 years
3. Patients with moderate to severe disease activity (DAS28>3.2)
4. Patients who have failed to respond to initial Methotrexate monotherapy

Exclusion Criteria:

1. End stage disease (deformed fixed joints)
2. Patients with vasculitis, extra-articular features like interstitial lung disease8
3. Contraindications to DMARD therapy (Chronic Alcoholism, Chronic liver disease, Evidence of acute/chronic infection, Chronic kidney disease, Patients with leucopenia (<3.0×109/l), thrombocytopenia (<150×109/l), AST/ALT>2× upper normal value and creatinine clearance <30ml/minute )
4. Pregnant, lactating women ; patients (both men and women) of reproductive age group unwilling for contraceptive use who have not completed the family
5. Patients unable to come for regular follow up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vir S Negi, DM, Principal Investigator — Jawaharlal Institute of Postgraduate Medical Education & Research; Pooja Belani, MD, Study Chair — Jawaharlal Institute of Postgraduate Medical Education & Research
Locations (1):
- Department of Clinical Immunology , Jawaharlal Institute of Post graduate Medical Educationa and Research, Puducherry, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belani PJ, Kavadichanda CG, Negi VS. Comparison between leflunomide and sulfasalazine based triple therapy in methotrexate refractory rheumatoid arthritis: an open-label, non-inferiority randomized controlled trial. Rheumatol Int. 2022 May;42(5):771-782. doi: 10.1007/s00296-021-04994-1. Epub 2021 Sep 29. PMID 34586472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were enrolled from OPD (outdoor patient department) of Rheumatology clinic of JIPMER , from September 2016 to March 2018
Period: Overall Study
Arm/Group | Group 1- MTX+LEF+HCQ | Group 2- MTX+SSZ+HCQ
Started | 68 | 68
Completed | 59 | 61
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1- MTX+LEF+HCQ | Group 2- MTX+SSZ+HCQ | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Customized [Median (Inter-Quartile Range); unit: years] — All patients above 18 years age, satisfying inclusion criteria were included
  years
    Age (years) | 39 [31 to 47] | 42 [29 to 46] | 40 [30 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 64 | 128
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease duration (months) [Median (Inter-Quartile Range); unit: months] | 12 [6 to 24] | 18 [6 to 24] | 15 [6 to 24]
Rheumatoid factor positivity [Count of Participants; unit: Participants] — Rheumatoid factor was evaluated by the Nephelometry method. A value of more than equal to 20IU/ml was considered positive
  Participants | 51 | 44 | 95
Anti- cyclic citrullinated peptide antibody [Count of Participants; unit: Participants] | 51 | 54 | 105
DAS28ESR [Median (Inter-Quartile Range); unit: units on a scale] — Full form : Disease activity score 28 joint ESR Measure of disease activity. Calculated from tender joint count, swollen joint count, patient VAS for global health and ESR.
  score ranges from 0 to 9.3 Higher score indicates higher disease activity
  units on a scale | 4.3 [4.1 to 5] | 4.2 [3.9 to 4.5] | 4.2 [4.1 to 4.7]
Tender joint count (TJ28) [Median (Inter-Quartile Range); unit: tender joints] — Includes the number of tender joints by palpation (includes all joints of both hands except distal interphalangeal joints, both elbows, both shoulders and both knees) Ranges from 0 to 28.
  tender joints | 4 [2 to 6] | 4 [2 to 5] | 4 [3 to 6]
Swollen joint count (SJ28) [Median (Inter-Quartile Range); unit: swollen joints] — Includes the number of joints that are swollen as per the examing physician. includes all joints of both hands (except distal interphalangeal joints), both wrists, elbows , shoulders and knees. Ranges from 0 to 28
  swollen joints | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Baseline ESR (mm at the end of 1 hour) [Median (Inter-Quartile Range); unit: millimeter (mm)] — ESR was measured using Westergren tube. The value ranges from 0 to 200 millimeters (mm).
  millimeter (mm) | 45 [35 to 52] | 40 [35 to 45] | 45 [35 to 50]
Early morning stiffness (EMS) (minutes) [Median (Inter-Quartile Range); unit: minutes] | 60 [30 to 60] | 60 [30 to 60] | 60 [30 to 60]
patient VAS global health [Median (Inter-Quartile Range); unit: units on a scale] — Value ranges from 0 to 100. Higher value indicates worse disease for patient overall health
  units on a scale | 20 [20 to 30] | 20 [10 to 30] | 20 [10 to 30]
Indian Health assessment questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Value ranges from 0 to 3 (calculated from 12 questions) where higher score indicates worse disease
  units on a scale | 1.9 [1.5 to 2.2] | 1.75 [1.2 to 2.5] | 1.8 [1.4 to 2.2]
Ultrasound7 score (US7 score) [Median (Inter-Quartile Range); unit: units on a scale] — Calculated from ultrasound assessment of 7 joints. Calcutes for disease activity (synovitis and effusion) and damage (erosions) using grey scale and power doppler Ranges from 0 to 108 Higher score indicates higher disease activity
  units on a scale | 3.5 [0 to 6] | 4 [0 to 4.5] | 4 [0 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Good EULAR Response at the End of 12 Weeks
Description: EULAR response criteria for Rheumatoid arthritis includes- estimation of DAS 28 ESR, that includes-
  1. Tender joint count 28
  2. Swollen joint count 28
  3. ESR
  4. Patient global assessment of health
Time Frame: 12 weeks
Population: Analysis was done by intention to treat
Measure: Number; unit: participants
Arm/Group | Group 1- MTX+LEF+HCQ | Group 2- MTX+SSZ+HCQ
Number analyzed (Participants) | 68 | 68
participants | 40 | 37

2. Secondary Outcome: Disease Activity as Per Ultrasound-7 (US-7) Score
Description: Ultrasound 7 score (US-7) Calculates ultrasound score in 7 joints using greyscale and power doppler to evaluate for disease activity (synovitis, tenosynovitis) and damage (erosions) Score minimum value= 0 Maximum value = 108 Higher score indicates worse disease
Time Frame: 12 weeks
Population: intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1- MTX+LEF+HCQ | Group 2- MTX+SSZ+HCQ
Number analyzed (Participants) | 68 | 68
units on a scale | 3.5 [0 to 6] | 4 [0 to 4.5]

3. Secondary Outcome: Number of Participants With Adverse Drug Reactions
Description: Infections, transaminitis, nausea, vomiting, derranged renal function tests etc
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1- MTX+LEF+HCQ | Group 2- MTX+SSZ+HCQ
Number analyzed (Participants) | 68 | 68
Participants
  Total number of any adverse events | 15 | 21
  Serious adverse events | 0 | 0
  Any gastrointestinal adverse reaction | 11 | 16
  Nausea | 4 | 6
  Diarrhea | 1 | 1
  Switch to parenteral Methotrexate | 5 | 14
  Raised liver enzymes > 2 times upper limit normal | 1 | 1
  Herpes labialis | 0 | 2
  upper respiratory tract infection | 5 | 5
  urinary tract infection | 1 | 0
  Hypertension | 1 | 0
  hairfall | 2 | 2
  Cytopenia | 0 | 0

4. Secondary Outcome: Indian Health Assessment Questionnaire (iHAQ)
Description: Indian version of Health assessment Questionnaire (iHAQ) Comprises of 12 questions relating to functional activity iHAQ score ranges from 0 to 3 (minimum 0, maximum 3) Higher scores indicate more disability
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group 1- MTX+LEF+HCQ | Group 2- MTX+SSZ+HCQ
Number analyzed (Participants) | 68 | 68
score on a scale | 0.7 [0.4 to 1] | 0.5 [0.07 to 1.3]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events were assessed for at each patient visit (clinical assessment and laboratory reports). Also, patients were given the contact number of researcher so that they can contact in case of any adverse reaction.
Arm/Group | Group 1- MTX+LEF+HCQ | Group 2- MTX+SSZ+HCQ
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 15/68 | 21/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- MTX+LEF+HCQ (N=68) | Group 2- MTX+SSZ+HCQ (N=68)
Gastrointestinal adverse events (Gastrointestinal disorders) | 11 (11) | 16 (16) — Includes nausea, vomiting, abdominal pain and diarrhea
infections (Infections and infestations) | 6 (6) | 7 (7) — Any infection during study period was noted
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hairfall (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Raised liver enzymes (Hepatobiliary disorders) | 1 (1) | 1 (1) — Liver enzymes > 2 times upper limit normal
Switch to parenteral Methotrexate (Product Issues) | 5 (5) | 14 (14) — Patients intolerant to Methotrexate were switched to parenteral form as per study protocol

LIMITATIONS AND CAVEATS:
Early termination resulted in enrollment of 136 patients instead of 140 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT02930343/Prot_SAP_ICF_000.pdf